CLINICAL TRIAL: NCT03712995
Title: Reconstruction of Upper Eyelid Defects Secondary to Malignant Tumors With a Newly Modified Cutler-Beard Technique With Tarsoconjunctival Graft
Brief Title: Reconstruction of Upper Eyelid With a Newly Modified Cutler-Beard Technique With Tarsoconjunctival Graf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RUE-2018
Record Dates: First submitted 2018-10-10; First posted 2018-10-19 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-10

CONDITIONS: Reconstructive Surgical Procedure
Keywords: Cutler-Beard; tarsoconjunctival graft; upper eyelid
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Intervention Model Description: Retrospective review of charts of the patients enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cutler-Beard modified with graft (Experimental): Reconstruction of Upper Eyelid With a Newly Modified Cutler-Beard Technique With Tarsoconjunctival Graf
  Interventions: Procedure: 'Cutler-Beard modified with graft'

INTERVENTIONS:
Procedure: 'Cutler-Beard modified with graft' — A tarsoconjunctival graft was harvested from the contralateral upper eyelid, with an extra 3 mm of conjunctiva from the superior edge of tarsus and was attached to the upper eyelid defect, differently than previously described.
  Other Names: Modified Cutler-Beard technique with tarsoconjunctival graft

SUMMARY:
To study the results of a modified Cutler-Beard technique , using a contralateral tarsoconjunctival graft, in patients who underwent excision of large malignant tumors of the upper eyelid

DETAILED DESCRIPTION:
A tarsoconjunctival graft was harvested from the contralateral upper eyelid, with an extra 3 mm of conjunctiva from the superior edge of tarsus and was attached to the upper eyelid defect, differently than previously described.

Functional, cosmetic outcomes and postoperative complications were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Upper eyelid defect after tumor resection

Exclusion Criteria:

* previous surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Eyelid retraction | 42 months
  Upper eyelid retraction in mm

SECONDARY OUTCOMES:
Retraction of the donor lower eyelid | 42 months
  Lower eyelid retraction in mm
Lagophthalmos | 42 months
  Excessive aperture of the eyelids, in mm
Lid margin stability | 42 months
  in mm
Eyelid status | 42 months
  Number of complications, being 0 the best result

OTHER OUTCOMES:
Symptoms of the patients | 42 months
  Number of symptoms referred by the patient, being 0 the best result

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Mencía-Gutiérrez, MD, Study Chair — Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Publication of the results in a journal